CLINICAL TRIAL: NCT01419236
Title: A Randomized, Double-Blind, Placebo-Controlled, Proof-of-Concept Study to Explore the Impact of Testosterone Solution 2% on Symptoms of Ejaculatory Dysfunction in Men With Testosterone Deficiency
Brief Title: A Study of Ejaculatory Dysfunction in Men With Low Testosterone Levels
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13981; I5E-MC-TSAB (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Results first posted 2014-12-19 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Ejaculatory Dysfunction; Hypogonadism
Keywords: Ejaculatory Dysfunction; Orgasmic Dysfunction; Sexual Dysfunction; Climax Dysfunction; Erectile Dysfunction; Impotence; Hypogonadism; Low testosterone; Low t
MeSH Terms: conditions — Ejaculatory Dysfunction; Hypogonadism; Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological; Erectile Dysfunction | interventions — Testosterone Propionate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Testosterone Solution 2% 60 milligrams (mg) (Experimental): Testosterone Solution 2% 60 mg applied topically once daily with possible 1-time titration to 30 milligrams per day (mg/day) or 90 mg/day for 16 weeks
  Interventions: Drug: Testosterone Solution 2%
- Placebo (Placebo Comparator): Placebo solution applied topically once daily for 16 weeks
  Interventions: Drug: Placebo Solution

INTERVENTIONS:
Drug: Testosterone Solution 2% — Administered topically
  Other Names: Axiron; LY900011
  Arms: Testosterone Solution 2% 60 milligrams (mg)
Drug: Placebo Solution — Administered topically
  Arms: Placebo

SUMMARY:
The purpose of this study is to see if testosterone solution 2% can impact symptoms of ejaculatory dysfunction in men with low testosterone.

ELIGIBILITY:
Inclusion Criteria:

* Total testosterone level <10.4 nanomoles per liter (nmol/L) [300 nanograms per deciliter (ng/dL)] at screening
* Presents with 1 or more of the following symptom(s) of ejaculatory dysfunction: delayed ejaculation, anejaculation, decreased force of ejaculation, or decreased ejaculatory volume, as determined by investigator assessment
* Prostate-Specific Antigen (PSA) <4 nanograms per milliliter (ng/mL) at screening

Exclusion Criteria:

* Sexual partner who is or becomes pregnant at any time during the study
* Premature ejaculation as determined by investigator assessment
* Currently receiving testosterone replacement therapy or have a history of insufficient response to testosterone replacement therapy for ejaculatory dysfunction symptoms
* Currently receiving treatment with cancer chemotherapy or antiandrogens
* History of use of estrogenizing agents
* Current use of warfarin
* History of selective serotonin reuptake inhibitor (SSRI) and/or serotonin-norepinephrine reuptake inhibitor (SNRI) treatment in the 6 months prior to screening
* History of frequent opioid use within 30 days prior to screening, with exception of treatment for chronic pain as determined by investigator.
* Body Mass Index (BMI) >35 kilograms per square meter (kg/m^2) at screening
* Significant peripheral neuropathy affecting erectile, ejaculatory, or orgasmic function
* Hematocrit ≥50% at screening
* Exhibit systolic blood pressure >170 millimeters of mercury (mm Hg) or <90 mm Hg or diastolic blood pressure >100 mm Hg or <50 mm Hg at screening (if stress is suspected, retest under basal conditions at screening), or have history of malignant hypertension
* History of any of the following coronary conditions within 90 days of screening: myocardial infarction, coronary artery bypass graft surgery, percutaneous coronary intervention (for example, angioplasty or stent placement)
* Known or suspected carcinoma (or history of carcinoma) of the prostate or suspicious nodules on digital rectal exam at screening
* Known or suspected breast cancer (or history of breast cancer) or other active cancer (with the exception of nonmelanotic skin cancer)

Min Age: 26 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2011-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Los Angeles, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New Orleans, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brookline, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Great Neck, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., New York, New York
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec, Quebec, Canada

REFERENCES:
- [Derived] Lee H, Hwang EC, Oh CK, Lee S, Yu HS, Lim JS, Kim HW, Walsh T, Kim MH, Jung JH, Dahm P. Testosterone replacement in men with sexual dysfunction. Cochrane Database Syst Rev. 2024 Jan 15;1(1):CD013071. doi: 10.1002/14651858.CD013071.pub2. PMID 38224135
- [Derived] Paduch DA, Polzer PK, Ni X, Basaria S. Testosterone Replacement in Androgen-Deficient Men With Ejaculatory Dysfunction: A Randomized Controlled Trial. J Clin Endocrinol Metab. 2015 Aug;100(8):2956-62. doi: 10.1210/jc.2014-4434. Epub 2015 Jul 9. PMID 26158605

RESULTS

PARTICIPANT FLOW:
Groups:
- Testosterone Solution 2%: Testosterone solution 2% [60 milligrams (mg) applied topically once daily with a potential 1-time titration to 30 milligrams per day (mg/day) or 90 mg/day] for 16 weeks.
Period: Overall Study
Arm/Group | Testosterone Solution 2% | Placebo
Started | 36 | 40
Received at Least 1 Dose of Study Drug | 35 | 39
Completed | 31 | 35
Not Completed | 5 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 1 | 4
Not completed — Entry Criteria Not Met | 1 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Testosterone Solution 2%: Testosterone solution 2% [60 mg applied topically once daily with a potential 1-time titration to 30 mg/day or 90 mg/day] for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Testosterone Solution 2% | Placebo | Total
Number analyzed (Participants) | 36 | 40 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.4 (9.83) | 52.7 (9.34) | 50.7 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 36 | 40 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 14
  Not Hispanic or Latino | 26 | 36 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 23 | 28 | 51
  More than one race | 0 | 3 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60
  Canada | 3 | 7 | 10
  Mexico | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Male Sexual Health Questionnaire-Ejaculatory Dysfunction-Short Form (MSHQ-EjD-SF) Ejaculatory Function Score at 16 Weeks
Description: MSHQ-EjD-SF: 4 item, self-reported questionnaire assessing ejaculatory dysfunction. MSHQ-EjD-SF Ejaculatory Function Score: sum of scores for questions (Q)1 through Q3 about frequency and strength of ejaculations and volume of ejaculate for sexual activity attempts during past month. Ejaculation frequency was rated 1 (could not ejaculate) to 5 (all the time); strength and volume from 0 (could not ejaculate) to 5 (as strong/much as it always has been). Total Ejaculatory Function Score ranged from 1 to 15. Least-squares (LS) mean of change from baseline calculated using repeated measures mixed-effects model (MMRM) including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level [≥200 nanograms per deciliter (ng/dL) versus (vs.) <200 ng/dL], baseline erectile dysfunction (ED) severity (normal, mild, moderate, severe), and centered baseline ejaculatory function score as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: Randomized participants who received at least 1 dose of study drug and completed the MSHQ-EjD-SF questionnaire at least once post-baseline.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
units on a scale | 3.61 (0.88) | 2.95 (0.81)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.380, Mixed Models Repeated Measure Analysis; LS Mean Difference = 0.66, 90% CI 2-sided [-0.59 to 1.91]

2. Secondary Outcome: Change From Baseline in Ejaculate Volume at 16 Weeks
Description: The change from baseline in ejaculate volume was determined by actual measurement of semen volume in milliliters (mL). LS mean of change from baseline was calculated using MMRM including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level (≥200 ng/dL vs. <200 ng/dL), baseline ED severity (normal, mild, moderate, severe), and centered baseline ejaculatory volume as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mL
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
mL | -0.12 (0.23) | 0.32 (0.21)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.164, Mixed Models Repeated Measures Analysis; LS Mean Difference = -0.44, 90% CI 2-sided [-0.96 to 0.08]

3. Secondary Outcome: Change From Baseline in Sexual Activity Log: Perceived Volume of Ejaculate at 16 Weeks
Description: The sexual activity log was used by study participants to document ejaculatory functioning and orgasmic pleasure for each sexual activity attempt over 4 weeks. Ejaculatory functioning included perceived volume of ejaculate, perceived force of ejaculation, delayed ejaculation, and frequency. Reported is the perceived volume of ejaculate rated from 0 (no ejaculate) to 10 (high volume of ejaculate). LS mean of change from baseline was calculated using MMRM including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level (≥200 ng/dL vs. <200 ng/dL), baseline ED severity (normal, mild, moderate, severe), and centered baseline ejaculatory volume as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
units on a scale | 1.85 (0.31) | 1.43 (0.30)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.342, Mixed Models Repeated Measure Analysis; LS Mean Difference = 0.42, 90% CI 2-sided [-0.31 to 1.15]

4. Secondary Outcome: Change From Baseline in Sexual Activity Log: Perceived Force of Ejaculation at 16 Weeks
Description: The sexual activity log was used by study participants to document ejaculatory functioning and orgasmic pleasure for each sexual activity attempt over 4 weeks. Ejaculatory functioning included perceived volume of ejaculate, perceived force of ejaculation, delayed ejaculation, and frequency. Reported is the perceived force of ejaculation rated from 0 (could not ejaculate) to 10 (strong ejaculation). LS mean of change from baseline was calculated using MMRM including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level (≥200 ng/dL vs. <200 ng/dL), baseline ED severity (normal, mild, moderate, severe), and centered baseline perceived force of ejaculation as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
units on a scale | 2.28 (0.32) | 1.47 (0.31)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.079, Mixed Models Repeated Measure Analysis; LS Mean Difference = 0.81, 90% CI 2-sided [0.05 to 1.57]

5. Secondary Outcome: Change From Baseline in Sexual Activity Log: Delayed Ejaculation at 16 Weeks
Description: The sexual activity log was used by study participants to document ejaculatory functioning and orgasmic pleasure for each sexual activity attempt over 4 weeks. Ejaculatory functioning included perceived volume of ejaculate, perceived force of ejaculation, delayed ejaculation, and frequency. Reported is delayed ejaculation rated from 0 (did not ejaculate) to 10 (optimal/best ejaculate time). LS mean of change from baseline was calculated using MMRM including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level (≥200 ng/dL vs. <200 ng/dL), baseline ED severity (normal, mild, moderate, severe), and centered baseline delayed ejaculation as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
units on a scale | 1.68 (0.34) | 1.38 (0.33)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.535, Mixed Models Repeated Measure Analysis; LS Mean Difference = 0.30, 90% CI 2-sided [-0.50 to 1.10]

6. Secondary Outcome: Change From Baseline in Sexual Activity Log: Frequency of Sexual Attempts at 16 Weeks
Description: The sexual activity log was used by study participants to document ejaculatory functioning and orgasmic pleasure for each sexual activity attempt over 4 weeks. Ejaculatory functioning included perceived volume of ejaculate, perceived force of ejaculation, delayed ejaculation, and frequency. Reported is the change from baseline number of sexual attempts at 16 weeks. LS mean of change from baseline was calculated using an analysis of covariance (ANCOVA) including treatment group, region, baseline total testosterone level, baseline ED severity (normal, mild, moderate, severe) as fixed effects, and centered baseline as a covariate.
Time Frame: Baseline, up to 16 weeks
Population: Randomized participants who received at least 1 dose of study drug and completed the MSHQ-EjD-SF questionnaire at least once post-baseline; Last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: sexual attempts
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
sexual attempts | 0.89 (0.53) | -0.14 (0.51)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.172, ANCOVA; LS Mean Difference = 1.03, 90% CI 2-sided [-0.22 to 2.27]

7. Secondary Outcome: Change From Baseline in Sexual Activity Log: Orgasmic Pleasure at 16 Weeks
Description: The sexual activity log was used by study participants to document ejaculatory functioning and orgasmic pleasure for each sexual activity attempt over 4 weeks. Reported is orgasmic pleasure rated from 0 (no pleasure) to 10 (excellent). LS mean of change from baseline was calculated using MMRM including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level (≥200 ng/dL vs. <200 ng/dL), baseline ED severity (normal, mild, moderate, severe), and centered baseline orgasmic pleasure as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
units on a scale | 1.37 (0.31) | 1.05 (0.30)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.473, Mixed Models Repeated Measure Analysis; LS Mean Difference = 0.32, 90% CI 2-sided [-0.41 to 1.04]

8. Secondary Outcome: Change From Baseline in the International Index of Erectile Function (IIEF)-Orgasmic Function Domain Score at 16 Weeks
Description: IIEF: 15 item, self-reported questionnaire assessing overall erectile function and satisfaction during past month. Orgasmic Function Domain Score: sum of IIEF scores for Q9 and Q10. In Q9, participants (pts) identified how often they ejaculated when having sexual stimulation or intercourse. In Q10, pts identified how often they had a feeling of an orgasm with or without ejaculation when having sexual stimulation or intercourse. For each Q, scores ranged from 0 (no sexual stimulation or intercourse), 1 (almost never or never) to 5 (almost always or always). Total Orgasmic Function Domain Scores ranged from 0 to 10. LS mean of change from baseline calculated using MMRM including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level (≥200 ng/dL vs. <200 ng/dL), baseline ED severity (normal, mild, moderate, severe), and centered baseline Orgasmic Function Domain Score as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
units on a scale | 1.21 (0.42) | 1.29 (0.38)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.885, Mixed Models Repeated Measure Analysis; LS Mean Difference = -0.08, 90% CI 2-sided [-1.03 to 0.87]

9. Secondary Outcome: Change From Baseline in MSHQ-EjD-SF Bother/Satisfaction Score at 16 Weeks
Description: The MSHQ-EjD-SF was a 4 item, self-reported questionnaire used for the assessment of EjD during the past month. The MSHQ-EjD-SF Bother/Satisfaction Score was based on Q4: "If you have had any ejaculation difficulties or have been unable to ejaculate, have you been bothered by this?" Scores ranged from 0 (no problem with ejaculation), 1 (not at all bothered) to 5 (extremely bothered). LS mean of change from baseline was calculated using MMRM including treatment, visit, treatment-by-visit interaction, region, baseline total testosterone level (≥200 ng/dL vs. <200 ng/dL), baseline ED severity (normal, mild, moderate, severe), and centered baseline Bother/Satisfaction Score as fixed effects, and unstructured covariance structure for modeling correlation.
Time Frame: Baseline, 16 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Testosterone Solution 2% | Placebo
Number analyzed (Participants) | 35 | 38
units on a scale | -1.65 (0.39) | -1.62 (0.36)
Statistical Analysis 1: Comparison: Testosterone Solution 2% vs Placebo; Test type: Superiority or Other; p = 0.938, Mixed Models Repeated Measure Analysis; LS Mean Difference = -0.03, 90% CI 2-sided [-0.61 to 0.55]

ADVERSE EVENTS:
Arm/Group | Testosterone Solution 2% | Placebo
Serious Adverse Events (participants affected / at risk) | 0/36 | 2/40
Other Adverse Events (participants affected / at risk) | 18/36 | 14/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Solution 2% (N=36) | Placebo (N=40)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Solution 2% (N=36) | Placebo (N=40)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Application site erythema (General disorders) | 1 (2) | 1 (1)
Application site pain (General disorders) | 1 (1) | 0 (0)
Application site paraesthesia (General disorders) | 0 (0) | 1 (1)
Application site pruritus (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Axillary candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Scar (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 0 (0) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0)
Glycosylated haemoglobin increased (Investigations) | 0 (0) | 1 (1)
Haematocrit increased (Investigations) | 3 (3) | 0 (0)
Haemoglobin increased (Investigations) | 1 (1) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Emotional disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 1 (1)
Libido increased (Psychiatric disorders) | 1 (1) | 0 (0)
Mood swings (Psychiatric disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Gynaecomastia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Testicular hypertrophy (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Skin neoplasm excision (Surgical and medical procedures) | 0 (0) | 1 (2)
Hot flush (Vascular disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days